CLINICAL TRIAL: NCT02117349
Title: A Phase 2, Randomized, Single-Blind, Controlled Trial of Topical Raplixa™ (Fibrin Sealant [Human]) in Intraoperative Surgical Hemostasis in a Pediatric Population
Brief Title: Topical Raplixa for Surgical Bleeding in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Non-safety device related issues
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FC-007
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Surgical Bleeding
Keywords: surgical hemostasis; bleeding; fibrin sealant; fibrinogen; thrombin; spray dried
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive; Gelatin Sponge, Absorbable; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Raplixa plus Gelfoam (Experimental): During a single predefined surgical procedure, participants receive the assigned treatment on an appropriate target bleeding site (TBS). The treatment is topically applied using 1 of the following 3 methods:
  * A thin layer of Raplixa is sprinkled directly from the vial onto the TBS, followed by application of Gelfoam.
  * A thin layer of Raplixa is sprayed onto the TBS using the RaplixaSpray device, followed by application of Gelfoam.
  * Raplixa is applied onto moistened Gelfoam which is then applied to the TBS.
  Manual pressure is applied over the treatments using sterile gauze. The amount of Raplixa and Gelfoam used is at the discretion of the investigator, within the maximum of two 1 gram (g) vials of Raplixa that are permitted for each participant.
  Thrombin-containing hemostats included in standard of care at the site are permitted as rescue therapy after the 5-minute time-to-hemostasis (TTH) evaluation.
  Interventions: Drug: Raplixa; Device: Gelfoam; Drug: Rescue treatment
- Gelfoam Only (Other): During a single predefined surgical procedure, participants receive the assigned treatment on an appropriate TBS. Gelfoam is cut to the appropriate size and applied topically, according to the manufacturer's package insert, followed by manual pressure using sterile gauze.
  Thrombin-containing hemostats included in standard of care at the site are permitted as rescue therapy after the 5-minute TTH evaluation, if necessary.
  Interventions: Device: Gelfoam; Drug: Rescue treatment

INTERVENTIONS:
Drug: Raplixa — Raplixa is a biological product approved for use in adults to help control bleeding from small blood vessels when standard surgical techniques, such as suture, ligature or cautery, are ineffective or impractical. When applied to a bleeding site, Raplixa is dissolved in the blood and a reaction starts between the fibrinogen and thrombin proteins. This results in the formation of blood clots to help stop the bleeding.
  Other Names: Fibrin Sealant [Human]; Fibrocaps
  Arms: Raplixa plus Gelfoam
Device: Gelfoam — Gelfoam Sterile Sponge is a medical device (USP, Pfizer) intended for application to bleeding surfaces as a hemostatic. It is a water-insoluble, off-white, nonelastic, porous, pliable product. It may be cut without fraying, used wet or dry, and is able to absorb many times its weight in blood and other fluids.
  Other Names: Gelfoam 50; Gelfoam 100
Drug: Rescue treatment — Thrombin-containing hemostats included in standard care at the site
  Other Names: Standard Care

SUMMARY:
The purpose of the study is to determine if Raplixa plus Gelfoam is better than Gelfoam alone in stopping mild to moderate bleeding in children having surgery.

ELIGIBILITY:
Before Surgery Inclusion Criteria:

* Was at least 36 weeks gestational age at birth (if an infant less than 6 months old) and is no older than 17 years at time of treatment
* Has a legal representative (parent or guardian) who signed an institutional review board (IRB)-approved informed consent document
* If at least 7 years old or appropriate age as defined by local regulations, may be required to sign an IRB-approved assent document
* Is scheduled to undergo one of the surgical procedures described in the protocol
* If female and of child-bearing potential, subject has negative pregnancy test on the day of surgery (baseline)
* If a sexually active male or female of reproductive potential, agrees to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits

During Surgery Inclusion Criteria:

* Has mild or moderate bleeding/oozing
* Has TBS surface area no more than 100 cm^2
* Has not received any whole blood, fresh frozen plasma (FFP), cryoprecipitate, or platelets within 24 hours prior to study drug (packed red blood cell (PRBC) transfusions are allowed)
* Had no complication during surgery other than bleeding which, in the opinion of the Investigator, may interfere with the assessment of efficacy or safety

Exclusion Criteria:

* Has any clinically significant laboratory or vital sign value, chronic disease state, or congenital coagulation disorder (eg, hemophilia A or B) that the investigator determines could interfere with the assessment of efficacy or pose a safety risk to the participant
* Is unwilling to receive blood products
* Has known antibodies or hypersensitivity to porcine gelatine, Raplixa or any of it's components, or other thrombin preparations or coagulation factors
* Has medical, social, or psychosocial factors that, in the opinion of the Investigator, could impact safety of the participant or compliance with study procedures, including protocol-defined limits on participating in other clinical studies

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (13):
- United States (13):
  - Arizona Burn Center at Maricopa Medical Center, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Shriners Hospital for Children, Sacramento, California
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - SGM Physician Research Consortium, LLC, Wayne, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Seattle Children's Hospital - PIN, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 87 planned participants, only 55 were randomized before the trial was terminated early due to device related (non-safety) issues
Groups:
- Raplixa Plus Gelfoam: Participants treated with Raplixa in addition to Gelfoam
- Gelfoam Alone: Participants treated only with Gelfoam
Period: Overall Study
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone
Started | 37 | 18
Intent-to-treat Population (All randomized participants (group based on random assignment)) | 37 | 18
Safety Population (Randomized participants exposed to study drug (group based on actual treatment received)) | 36 | 18
Modified Intent-to-treat (mITT) (Randomized participants who received assigned study treatment and had no major protocol violations) | 36 | 18
Completed | 34 | 17
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: modified Intent-to-treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Continuous [Median (Full Range); unit: years] | 6.6 [0.9 to 16.9] | 9.7 [2.7 to 17.8] | 6.9 [0.9 to 17.8]
Age, Customized [Count of Participants; unit: Participants] — Number of Participants in the mITT population for each Age Cohort
  Participants
    Age Cohorts: Cohort 1 = 11 to < 18 years | 13 | 9 | 22
    Age Cohorts: Cohort 2 = 2 to < 11 years | 19 | 9 | 28
    Age Cohorts: Cohort 3 = 6 months to < 2 years | 4 | 0 | 4
    Age Cohorts: Cohort 4 = Birth to < 6 months | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 21 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 22 | 10 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 26 | 9 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reached Hemostasis at the Target Bleeding Site (TBS) Within 4 Minutes
Description: Count of Participants who Reached Hemostasis at the TBS within 4 minutes of the first study drug application
Time Frame: within 4 minutes
Population: modified Intent to Treat (mITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone
Number analyzed (Participants) | 36 | 18
Participants | 30 | 5
Statistical Analysis 1: Comparison: Raplixa Plus Gelfoam vs Gelfoam Alone; Odds Ratio (OR) and Wald-based 95% Confidence intervals (CIs) are from logistic regression model comparing the response between treatment arms; Test type: Other; p = 0.0010, Regression, Logistic — Study was terminated early at 55 randomized subjects, therefore p-value is considered nominal; Odds Ratio (OR) = 42.8, 95% CI 2-sided [4.58 to 401.0]

2. Secondary Outcome: Number of Participants Who Reached Hemostasis at the TBS Within 5 Minutes
Description: Count of Participants who Reached Hemostasis at the TBS within 5 minutes of the first study drug application
Time Frame: within 5 minutes
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone
Number analyzed (Participants) | 36 | 18
Participants | 33 | 7

3. Secondary Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (TEAEs)
Description: Clinically significant changes in safety measures are recorded as adverse events. Participants with TEAEs that are deemed by the principal investigator or the independent data monitoring committee as possibly or definitely treatment-related (including device-related) are included in the count for this secondary outcome measure.
Time Frame: within 97 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone
Number analyzed (Participants) | 36 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: within 97 days
Description: All-cause mortality is reported in the Intent-to-treat population (37/18) to include one who was randomized, but died before treatment.
  Serious and Other Adverse events are reported in the Safety population (36/18), defined as randomized participants who were exposed to study drug (group based on actual treatment received).
Arm/Group | Raplixa Plus Gelfoam | Gelfoam Alone
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/36 | 1/18
Other Adverse Events (participants affected / at risk) | 0/36 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Raplixa Plus Gelfoam (N=36) | Gelfoam Alone (N=18)
Ascites (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Intussusception (Gastrointestinal disorders) | 1 | 1
Gastrointestinal norovirus (Infections and infestations) | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 1
Stoma site cellulitis (Infections and infestations) | 1 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Gastrointestinal stoma output abnormal (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT02117349/Prot_SAP_000.pdf